CLINICAL TRIAL: NCT02269137
Title: Assessment of Severity and Prognosis for Patients With Status Epileptics
Brief Title: Assessment of Severity and Prognosis for Patients With Status Epileptics(SE)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Xijing-49
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Status Epileptics
Keywords: status epileptics; prognosis; risk factor; outcome

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To characterize the functional outcomes and prognostic factors for convulsive status epilepticus (SE) and to further develop and validate a simple and practicable scoring system for outcome prediction.

DETAILED DESCRIPTION:
1. Retrospectively study all patients with convulsive SE treated between March, 2008, and November, 2014.
2. Develop a scoring system for outcome prediction.
3. Prospectively validate the predictive accuracy of the scoring system

ELIGIBILITY:
Inclusion Criteria:

* 30 min or more of (1) continuous clinical seizure activities or (2) recurrent seizure activities without recovery(returning to baseline)between seizures;
* clinical data is complete.

Exclusion Criteria:

* hypoglycemia SE;psychogenic SE;any other pseudo-SE

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with status epilepticus
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-03; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin scale | 3 months after discharge

SECONDARY OUTCOMES:
The modified Rankin scale | on discharge

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, MD, Study Director — The Department of Neurology, Xijing Hospital
Locations (1):
- The Department of Neurology, Xijing Hospital, Xi'an, Shaanxi, China